CLINICAL TRIAL: NCT03226769
Title: Prospective, Open-Label, Randomized, Proof of Concept Study Exploring Application of TrueTear™ for the Treatment of Meibomian Gland Disease
Brief Title: Safety and Efficacy of TrueTear™ for the Treatment of Meibomian Gland Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OCUN-023
Record Dates: First submitted 2017-07-20; First posted 2017-07-24 (Actual); Results first posted 2020-10-30 (Actual); Last update posted 2020-10-30 (Actual); Status verified 2020-10

CONDITIONS: Meibomian Glands; Dry Eye Syndromes
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Thermalon (Active Comparator): Participants received application of Thermalon dry eye compress on Days 0 and 7 followed by daily use as per label instructions.
  Interventions: Device: Thermalon Dry Eye Compress
- TrueTear™ (Experimental): Participants received TrueTear™ device intranasally for approximately 8 minutes on Day 0, for approximately 3 minutes on Day 7 followed by daily use of TrueTear™ per participant guide.
  Interventions: Device: TrueTear™

INTERVENTIONS:
Device: TrueTear™ — Intranasal application of TrueTear™ device for approximately 8 minutes at Day 0, for approximately 3 minutes at Day 7 and then daily use of TrueTear™ per participant guide.
  Arms: TrueTear™
Device: Thermalon Dry Eye Compress — Application of Thermalon Dry Eye Compress at Day 0, Day 7 and daily use as per label instructions.
  Arms: Thermalon

SUMMARY:
This study will compare the safety and efficacy of TrueTear™ to standardized moist heat compress (Thermalon® Dry Eye Compress) for the treatment of Meibomian Gland Disease (MGD).

ELIGIBILITY:
Inclusion Criteria:

* Dry eye disease or Meibomian Gland Disease as evaluated by Standard Participant Evaluation for Dryness (SPEED) score, Schirmer test, Tear film breakup time and other applicable objective measures at the Screening and Baseline Visits.
* Use of an artificial tear product, lid hygiene, omega-3 supplementation, antibiotics for the treatment of dry eye disease or Meibomian Gland Disease within one year of the Screening Visit.

Exclusion Criteria:

* Chronic or recurrent epistaxis, coagulation disorders or other conditions that may increase the risk of bleeding.
* History of nasal or sinus surgery.
* Vascularized polyp, deviated septum or severe nasal airway obstruction at the Screening visit.
* Intraocular and extraocular surgery in either eye within three months of the Screening Visit or refractive surgery within twelve months of the Screening Visit.
* Cardiac demand pacemaker, implanted defibrillator, or other active implanted metallic or active implanted electronic device in the head.

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2017-07-26 (Actual); Primary Completion 2017-12-12 (Actual); Study Completion 2017-12-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gail Torkildsen, Principal Investigator — mdlasik@comcast.net
Locations (1):
- Andover Eye Associates, Andover, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Thermalon | TrueTear™
Started | 29 | 28
Completed | 29 | 27
Not Completed | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Population: Intent-to-treat (ITT) population included all randomized participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Thermalon | TrueTear™ | Total
Number analyzed (Participants) | 29 | 28 | 57
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.2 (12.16) | 63.8 (13.91) | 63.5 (12.94)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 19 | 37
  Male | 11 | 9 | 20
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 2 | 2
  Not Hispanic or Latino | 29 | 26 | 55
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 0 | 2
  White | 27 | 28 | 55
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Meibomian Gland Dysfunction (MGD) Impact Questionnaire Score [Mean (Full Range); unit: score on a scale] — MGD impact questionnaire includes 10 questions about impacts participant may experience associated with MGD. Question/s (Qs) 1-6 were rated on a scale of 1=no difficulty to 5=lot of difficulty. Q7 was rated on scale of 1=never to 5=all the time. If participants did not experience particular impact, they chose 0=Not applicable (NA) for Qs 1-7. Q8 was rated on scale 0-4, where 0=no time at all to 4=lot of time, Qs 9-10 were rated on scale 0-4, with 0=not at all bothered to 4=very bothered. Higher scores represented greater impact. For additional scale information see Outcome Measure section.
  score on a scale
    Computer Usage | 2.3 [0 to 4] | 2.0 [0 to 4] | 2.1 [0 to 4]
    Reading | 2.7 [1 to 4] | 2.0 [1 to 5] | 2.3 [1 to 5]
    Leisure Activities | 2.5 [1 to 4] | 2.2 [1 to 5] | 2.3 [1 to 5]
    Social Activities | 1.4 [0 to 3] | 1.7 [0 to 4] | 1.5 [0 to 4]
    Driving | 2.0 [1 to 4] | 2.1 [1 to 4] | 2.0 [1 to 4]
    Outdoor Activities | 1.9 [0 to 5] | 1.6 [0 to 4] | 1.7 [0 to 5]
    Frequency of Outdoor Activities | 2.0 [0 to 4] | 1.8 [0 to 5] | 1.9 [0 to 5]
    Time Spent to Take Care of Eyes | 1.7 [0 to 3] | 1.4 [0 to 3] | 1.5 [0 to 3]
    Bothered With Amount of Time Taking Care of Eyes | 1.3 [0 to 4] | 0.9 [0 to 3] | 1.1 [0 to 4]
    Bothered by Appearance | 1.1 [0 to 4] | 1.2 [0 to 4] | 1.1 [0 to 4]
MGD Symptoms Questionnaire Score [Mean (Full Range); unit: score on a scale] — MGD symptom questionnaire included 11 questions about the symptoms the participant may experience associated with MGD. The participant was asked to rate how much they experienced certain MGD symptoms and the severity of the symptoms over the past 24 hours on a scale of 0 to 4, where 0 = not at all, 1 = a little, 2 = somewhat, 3=quite a bit, 4 = very. A higher score within each question represented increased severity of the indicated symptom. For additional scale information see Outcome Measure section.
  score on a scale
    Red Eyes | 1.3 [0 to 4] | 1.2 [0 to 3] | 1.2 [0 to 4]
    Blurred Vision | 1.4 [0 to 3] | 1.2 [0 to 3] | 1.3 [0 to 3]
    Dry Eyes | 2.6 [1 to 4] | 2.5 [1 to 4] | 2.5 [1 to 4]
    Itchy Eyes | 2.2 [1 to 4] | 1.6 [0 to 4] | 1.9 [0 to 4]
    Burning Eyes | 1.5 [0 to 4] | 1.5 [0 to 4] | 1.5 [0 to 4]
    Gritty Eyes | 2.0 [1 to 4] | 1.7 [0 to 4] | 1.8 [0 to 4]
    Painful Eyes | 1.0 [0 to 3] | 0.9 [0 to 3] | 0.9 [0 to 3]
    Watery Eyes | 1.3 [0 to 4] | 1.3 [0 to 4] | 1.3 [0 to 4]
    Swollen Eyelids | 0.6 [0 to 3] | 0.5 [0 to 2] | 0.5 [0 to 3]
    Red Eyelids | 0.9 [0 to 4] | 1.0 [0 to 4] | 0.9 [0 to 4]
    Crusty Eyelids | 1.0 [0 to 4] | 1.1 [0 to 4] | 1.0 [0 to 4]

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Meibomian Gland Dysfunction (MGD) Impact Questionnaire Score
Description: MGD impact questionnaire includes 10 questions about the impacts a participant may experience associated with MGD. Participants were asked to rate how much they have been affected by MGD symptoms in past 7 days. Question/s (Qs) 1-6 (computer usage, reading, leisure activities, social activities, driving and outdoor activities) were rated on a scale of 1=no difficulty to 5=a lot of difficulty. Q7 (frequency of outdoor activities) was rated on scale of 1=never to 5=all the time. If participants did not experience a particular impact, they chose 0=NA for Qs 1-7. Q8 (time spent to take care of eyes) was rated on scale 0-4, where 0=no time at all to 4=a lot of time, Qs 9-10 (bothered with amount of time taking care of eyes and bothered by appearance) were rated on scale 0-4, with 0=not at all bothered to 4=very bothered. Higher scores represented greater impact. A negative change from Baseline indicates improvement.
Time Frame: Baseline (Day 0) to Day 30
Population: ITT population included all randomized participants. Overall number of participants analyzed is the number of participants with data available for analyses.
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Thermalon | TrueTear™
Number analyzed (Participants) | 29 | 27
score on scale
  Computer Usage | -0.4 (0.86) | -0.3 (0.83)
  Reading | -0.4 (0.90) | -0.2 (0.79)
  Leisure Activities | -0.3 (0.89) | -0.4 (0.89)
  Social Activities | -0.2 (0.87) | -0.2 (0.79)
  Driving | -0.1 (0.92) | -0.2 (1.05)
  Outdoor Activities | -0.3 (0.81) | -0.1 (0.85)
  Frequency of Outdoor Activities | -0.2 (0.69) | -0.1 (0.83)
  Time Spent to Take Care of Eyes | -0.1 (0.83) | 0.1 (0.91)
  Bothered With Amount of Time Taking Care of Eyes | -0.4 (1.01) | 0.0 (1.09)
  Bothered by Appearance | -0.3 (0.77) | -0.1 (0.82)
Statistical Analysis 1: Comparison: Thermalon vs TrueTear™; Computer Usage; Test type: Other — The null hypothesis is that there is no difference between the two devices, TrueTear™ and Thermalon; p = 0.9788, Wilcoxon rank-sum test — Statistically significant (p < 0.05) and trending significant (p < 0.10) for within-group or between-group changes from baseline at Day 30. Between-group P-value was calculated using Wilcoxon rank-sum test
Statistical Analysis 2: Comparison: Thermalon vs TrueTear™; Reading; Test type: Other — The null hypothesis is that there is no difference between the two devices, TrueTear™ and Thermalon; p = 0.6571, Wilcoxon rank-sum test — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Thermalon vs TrueTear™; Leisure Activities; Test type: Other — The null hypothesis is that there is no difference between the two devices, TrueTear™ and Thermalon; p = 0.4710, Wilcoxon rank-sum test — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: Thermalon vs TrueTear™; Social Activities; Test type: Other — The null hypothesis is that there is no difference between the two devices, TrueTear™ and Thermalon; p = 0.7360, Wilcoxon rank-sum test — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 5: Comparison: Thermalon vs TrueTear™; Driving; Test type: Other — The null hypothesis is that there is no difference between the two devices, TrueTear™ and Thermalon; p = 0.4999, Wilcoxon rank-sum test — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 6: Comparison: Thermalon vs TrueTear™; Outdoor Activities; Test type: Other — The null hypothesis is that there is no difference between the two devices, TrueTear™ and Thermalon; p = 0.1159, Wilcoxon rank-sum test — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 7: Comparison: Thermalon vs TrueTear™; Frequency of Outdoor Activities; Test type: Other — The null hypothesis is that there is no difference between the two devices, TrueTear™ and Thermalon; p = 0.4567, Wilcoxon rank-sum test — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 8: Comparison: Thermalon vs TrueTear™; Time Spent to Take Care of Eyes; Test type: Other — The null hypothesis is that there is no difference between the two devices, TrueTear™ and Thermalon; p = 0.3439, Wilcoxon rank-sum test — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 9: Comparison: Thermalon vs TrueTear™; Bothered With Amount of Time Taking Care of Eyes; Test type: Other — The null hypothesis is that there is no difference between the two devices, TrueTear™ and Thermalon; p = 0.3331, Wilcoxon rank-sum test — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 10: Comparison: Thermalon vs TrueTear™; Bothered by Appearance; Test type: Other — The null hypothesis is that there is no difference between the two devices, TrueTear™ and Thermalon; p = 0.4774, Wilcoxon rank-sum test — [p-value comment as in outcome 1, analysis 1]

2. Primary Outcome: Change From Baseline in MGD Symptoms Questionnaire Score
Description: MGD symptom questionnaire included 11 questions about the symptoms the participant may experience associated with MGD. The participant was asked to rate how much they experienced certain MGD symptoms and the severity of the symptoms over the past 24 hours on a scale of 0 to 4, where 0 = not at all, 1 = a little, 2 = somewhat, 3=quite a bit, 4 = very. A higher score within each question represented increased severity of the indicated symptom. A negative change from baseline indicates improvement.
Time Frame: Baseline (Day 0) to Day 30
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Thermalon | TrueTear™
Number analyzed (Participants) | 29 | 27
score on a scale
  Red Eyes | -0.2 (0.76) | -0.1 (0.83)
  Blurred Vision | -0.2 (0.85) | -0.2 (0.80)
  Dry Eyes | -0.3 (1.04) | -0.5 (0.85)
  Itchy Eyes | -0.8 (1.23) | -0.3 (0.99)
  Burning Eyes | -0.2 (0.77) | -0.5 (0.89)
  Gritty Eyes | -0.2 (0.99) | -0.4 (0.88)
  Painful Eyes | -0.4 (0.87) | -0.1 (0.62)
  Watery Eyes | 0.0 (1.20) | -0.1 (0.75)
  Swollen Eyelids | 0.0 (0.93) | 0.3 (0.66)
  Red Eyelids | 0.0 (0.78) | -0.1 (0.46)
  Crusty Eyelids | 0.1 (0.75) | -0.4 (0.74)
Statistical Analysis 1: Comparison: Thermalon vs TrueTear™; Red Eyes; Test type: Other — The null hypothesis is that there is no difference between the two devices, TrueTear™ and Thermalon; p = 0.5457, Wilcoxon rank-sum test — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Thermalon vs TrueTear™; Blurred Vision; Test type: Other — The null hypothesis is that there is no difference between the two devices, TrueTear™ and Thermalon; p = 0.9786, Wilcoxon rank-sum test — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Thermalon vs TrueTear™; Dry Eyes; Test type: Other — The null hypothesis is that there is no difference between the two devices, TrueTear™ and Thermalon; p = 0.3894, Wilcoxon rank-sum test — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: Thermalon vs TrueTear™; Itchy Eyes; Test type: Other — The null hypothesis is that there is no difference between the two devices, TrueTear™ and Thermalon; p = 0.0591, Wilcoxon rank-sum test — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 5: Comparison: Thermalon vs TrueTear™; Burning Eyes; Test type: Other — The null hypothesis is that there is no difference between the two devices, TrueTear™ and Thermalon; p = 0.1818, Wilcoxon rank-sum test — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 6: Comparison: Thermalon vs TrueTear™; Gritty Eyes; Test type: Other — The null hypothesis is that there is no difference between the two devices, TrueTear™ and Thermalon; p = 0.4284, Wilcoxon rank-sum test — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 7: Comparison: Thermalon vs TrueTear™; Painful Eyes; Test type: Other — The null hypothesis is that there is no difference between the two devices, TrueTear™ and Thermalon; p = 0.1051, Wilcoxon rank-sum test — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 8: Comparison: Thermalon vs TrueTear™; Watery Eyes; Test type: Other — The null hypothesis is that there is no difference between the two devices, TrueTear™ and Thermalon; p = 0.7998, Wilcoxon rank-sum test — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 9: Comparison: Thermalon vs TrueTear™; Swollen Eyelids; Test type: Other — The null hypothesis is that there is no difference between the two devices, TrueTear™ and Thermalon; p = 0.1229, Wilcoxon rank-sum test — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 10: Comparison: Thermalon vs TrueTear™; Red Eyelids; Test type: Other — The null hypothesis is that there is no difference between the two devices, TrueTear™ and Thermalon; p = 0.3907, Wilcoxon rank-sum test — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 11: Comparison: Thermalon vs TrueTear™; Crusty Eyelids; Test type: Other — The null hypothesis is that there is no difference between the two devices, TrueTear™ and Thermalon; p = 0.0336, Wilcoxon rank-sum test — [p-value comment as in outcome 1, analysis 1]

ADVERSE EVENTS:
Time Frame: Up to Day 30
Arm/Group | Thermalon | TrueTear™
All-Cause Mortality (participants affected / at risk) | 0/29 | 0/28
Serious Adverse Events (participants affected / at risk) | 0/29 | 0/28
Other Adverse Events (participants affected / at risk) | 2/29 | 2/28
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Thermalon (N=29) | TrueTear™ (N=28)
Vision blurred (Eye disorders) | 2 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.

DOCUMENTS (2):
  • Statistical Analysis Plan (2018-09-25): https://cdn.clinicaltrials.gov/large-docs/69/NCT03226769/SAP_000.pdf
  • Study Protocol (2017-06-01): https://cdn.clinicaltrials.gov/large-docs/69/NCT03226769/Prot_001.pdf